CLINICAL TRIAL: NCT05950971
Title: Rhythm Control Versus Rate Control for New Onset Atrial Fibrillation After Non-cardiac Non-thoracic Surgery
Brief Title: Rhythm Control Versus Rate Control for New Onset Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment too slow, 1 over 6 months
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Postoperative NOAF
Record Dates: First submitted 2021-12-05; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation New Onset; Atrial Fibrillation Paroxysmal
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Diltiazem; esmolol

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rate control strategy group (Experimental): Patients are given diltiazem or esmolol to control heart rate less than 110/min.
  Interventions: Drug: Amiodarone, diltiazem or esmolol
- Rhythm control strategy group (Experimental): Patients are given amiodarone for conversion of cardiac rhythm to sinus rhythm.
  Interventions: Drug: Amiodarone, diltiazem or esmolol

INTERVENTIONS:
Drug: Amiodarone, diltiazem or esmolol — Intravenous continuous infusion after loading or bolus dose of amiodarone, diltiazem or esmolol.
  Other Names: herben

SUMMARY:
Adult patients who are diagnosed new onset atrial fibrillation with rapid ventricular response within 7 days after non-cardiac non-thoracic surgery are enrolled.

DETAILED DESCRIPTION:
After randomization, they are allocated to rhythm control strategy group or rate control strategy group. In rhythm control strategy group, patients are given amiodarone primarily for the purpose of sinus conversion of cardiac rhythm. In rate control strategy group, patients are given diltiazem or esmolol for the purpose of rate control. the rate of sinus conversion within 48 hours after treatment are compared.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Newly diagnosed atrial fibrillation or flutter
* Patients with atrial fibrillation or flutter that occurred within 7 days after non-cardiac non-thoracic surgery
* Atrial fibrillation or flutter with rapid ventricular response(HR ≥110/min)
* Patients without hemodynamic instability (MBP≥65mmHg with norepinephrine continuous infusion less than 5mcg/min or without vasopressor support)

Exclusion Criteria:

* Atrial fibrillation or flutter prolonged more than 48 hours without anticoagulation
* Patients who have decreased cardiac function or heart failure (EF <40%)
* Patients who have cardiac conduction disorder, QT prolongation(QTc ≥500ms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Rate of sinus conversion | within 48 hrs
  Rate of sinus conversion within 48 hours

SECONDARY OUTCOMES:
Time to first sinus conversion | during the same admission period
  Time to first sinus conversion
Recurrence of atrial fibrillation | during the same admission period
  Recurrence of atrial fibrillation during the same admission period

CONTACTS AND LOCATIONS:
Overall Officials: Hogeol Ryu, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No